CLINICAL TRIAL: NCT05267886
Title: CAPITAL DOREMI 2: Inotrope Versus Placebo Therapy for Cardiogenic Shock
Acronym: DOREMI-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210386
Record Dates: First submitted 2022-02-03; First posted 2022-03-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Shock, Cardiogenic
Keywords: cardiogenic; shock; inotrope
MeSH Terms: conditions — Shock, Cardiogenic; Shock | interventions — Dobutamine; Milrinone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel randomized control trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inotrope (Active Comparator): Participants randomized to receive the inotrope will be initiated on inotrope therapy at starting doses and titrated according to standard clinical care. During reassessment, the treating physicians will make a decision about adjustment of the inotrope dose (increase, maintain or decrease) based on hemodynamics, end-organ perfusion, vasopressor support and clinical exam. Dobutamine doses will be 2.5, 5.0, 7.5, 10 and >10 ug/kg/min and milrinone doses will be 0.125, 0.250, 0.375, 0.5 and >0.5 ug/kg/min. These dose stages are identical to those used in Capital Do-Re-Mi and reflect current standard of care.
  Interventions: Drug: Dobutamine; Drug: Milrinone
- Placebo (Placebo Comparator): Participants in the placebo arm will have an intravenous solution of 0.9% NaCl running at a standardized rate, comparable to the infusion rate of the inotrope arm.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dobutamine — Dobutamine administered according to its clinical dose stage for cardiogenic shock
  Other Names: Dobutrex, Inotrex
  Arms: Inotrope
Drug: Milrinone — Milrinone administered according to its clinical dose stage for cardiogenic shock
  Arms: Inotrope
Drug: Normal Saline — Normal saline running at a standardized rate
  Arms: Placebo

SUMMARY:
The investigators are interested in determining if there is a meaningful benefit from the use of medications purported to increase the pumping function of the heart (i.e. inotropes) among critically ill patients admitted to the Cardiac Intensive Care Unit (CICU). To do this, the investigators will conduct a multi-centre, double blind, randomized control trial with patients who are deemed to require these medications by their treating physician to one of the two most commonly used agents in Canada (Milrinone or Dobutamine) or placebo. Each patient will be closely monitored by their healthcare team. The dose of medication will be adjusted according to each patients' clinical status. After 12 hours, the participants will move to open label treatment and any continued use of inotropes will be at the discretion of their treating physician.

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is a state of inadequate end-organ perfusion due to cardiac dysfunction. Acute myocardial infarction (AMI) remains the most prevalent cause of CS, with mortality reaching upwards of 40% despite advances in emergent revascularization and accelerating use of mechanical circulatory support devices. International guidelines support the use of vasopressors and inotropes as a mainstay of medical therapy among this cohort of critically ill patients. Recently, the first head-to-head prospective randomized trial (CAPITAL DOREMI) comparing milrinone and dobutamine in a cohort of CS participants was performed and found no difference between agents.

There is a signal of harm associated with the use of inotropes in both acute, decompensated heart failure and in the longitudinal management of chronic heart failure. Inotrope use has also been associated with longer ICU and in-hospital length of stay, as well as higher in-hospital mortality. A recent network meta-analysis on treatment strategies in CS and found that while milrinone and dobutamine may reduce the risk of mortality compared to placebo, the evidence is of low certainty and the wide confidence intervals do not rule out the possibility of harm.

Despite their frequent use in the management of patients with CS, it remains unknown if inotropes are needed to augment successful initial resuscitation, reduce morbidity and mortality, or if they cause potential harm in this already critically ill patient population.

This study is a multi-centre, double blind, randomized controlled trial designed to examine the efficacy and safety of inotrope therapy against placebo in the initial resuscitation of SCAI class C to D cardiogenic shock. Consecutive patients admitted to an intensive care unit will be identified by the treating medical team as requiring new initiation of inotrope therapy for CS. All decisions to initiate inotrope therapy will be made by the primary care team with no involvement from the research team. The study hypothesis is that inotrope therapy will lead to an overall improvement in the primary outcome as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age admitted to an intensive care unit
* SCAI class C or D cardiogenic shock

Exclusion Criteria:

* Unwilling or unable to obtain informed consent by the participant or substitute decision maker
* Patients who are currently pregnant or breast-feeding
* Patients presenting with an out-of-hospital cardiac arrest (OHCA)
* Administration of milrinone or dobutamine in the 24 hours preceding anticipated randomization
* Severe obstructive valvular lesions, including aortic stenosis and/or mitral stenosis
* Dynamic left ventricular outflow tract obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2022-03-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary composite outcome | Through duration of hospitalization, up to 12 weeks following admission
  The primary outcome will be a composite of:
  1. All-cause mortality during the hospitalization
  2. Measured within the first 12 hours of starting the study intervention, any of:
     1. Sustained hypotension (mean arterial pressure ≤55mmHg) or sustained requirement of high dose vasopressors (norepinephrine >0.2 mcg/kg/min or norepinephrine 0.2 mcg/kg/min plus any additional agent) with any escalation in dose from time of randomization, for >/= 60 minutes
     2. Lactate greater than 3.5 mmol/L at 6 hours or thereafter
     3. Need for mechanical circulatory support device
     4. Atrial or ventricular arrhythmia leading to emergent electrical cardioversion
     5. Resuscitated cardiac arrest

SECONDARY OUTCOMES:
All-cause in-hospital mortality | Through duration of hospitalization, up to 12 weeks following admission
  Death resulting from any cause during hospitalization
Renal failure requiring new initiation of renal replacement therapy | Through duration of hospitalization, up to 12 weeks following admission
  Requiring new initiation of renal replacement therapy
Need for cardiac transplant or mechanical circulatory support | Through duration of hospitalization, up to 12 weeks following admission
  Identification of needing a cardiac transplant or mechanical circulatory support
Atrial or ventricular arrhythmia leading to emergent electrical cardioversion | Through duration of hospitalization, up to 12 weeks following admission
  Requiring emergent electrical cardioversion for atrial or ventricular arrhythmia
Resuscitated cardiac arrest | Through duration of hospitalization, up to 12 weeks following admission
  Cardiopulmonary arrest requiring chest compressions and/or defibrillation with successful return of spontaneous circulation (ROSC)
Non-fatal myocardial infarction | Through duration of hospitalization, up to 12 weeks following admission
  Non-fatal myocardial infarction
Stroke or transient ischemic attack | Through duration of hospitalization, up to 12 weeks following admission
  Defined as an episode of focal or global neurological deficit as diagnosed by a neurologist

OTHER OUTCOMES:
Need for non-invasive or invasive mechanical ventilation | Through duration of hospitalization, up to 12 weeks following admission
  Need for non-invasive or invasive mechanical ventilation after randomization
Arrhythmia requiring pharmacologic intervention | Through duration of hospitalization, up to 12 weeks following admission
  Atrial or ventricular arrhythmias requiring initiation of pharmacologic intervention (intravenous or oral anti-arrhythmic therapy)
Acute kidney injury | Through duration of hospitalization, up to 12 weeks following admission
  Acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Mathew, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (3):
- Mayo Clinic, Rochester, Minnesota, United States
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The study data, protocol, SAP, ICF, and CSR will be made available at study completion/publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study completion
Access Criteria: The above will be made publicly available